CLINICAL TRIAL: NCT05135689
Title: Medico-social Description of Seniors Living With HIV, Associated With a Qualitative Survey on Their Care in the Paris Region Structures
Acronym: VIAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A01097-34
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: HIV-positive
Keywords: HIV-positive; Serophobia
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is part of a national vision to fight against serophobia and support society towards more ethical and benevolent practices vis-à-vis aging and specific populations.

The main objective of this study is to assess over the past five years the prevalence of people living with the Human Immunodeficiency Virus (HIV) aged 60 years and over and its evolution within the Paris Region medico-social structures

DETAILED DESCRIPTION:
The aim objective of this study is to identify patients living with the Human Immunodeficiency Virus (HIV) in medical and social strutures in Île-de-France, in order to question them, in particular about their life courses and how they are treated and supported now. This study also query family caregivers of seropositive seniors and profiessional caregivers.

This trial is designed in two parts:

* The one consists to quantify and describe patient's clinical and social profil: Age, sex, authonomy level, medical data related to HIV infoection, Chronic deseases, social and economic data will be collected at 5 and 3 years before inclusion, at inclusion, at 1 and 2 yeans after inclusion
* Then a second qualitative part which allow to query seropositive patients about their fagility and comorbidities, and to identify the impact of these on their life and social relation.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* HIV-positive, regardless of strain or age of infection,
* Orally expressing his non-opposition to his participation in the study and documented in the medical file by investigator,
* Follow-up, placed and / or treated in one of the centers concerned by the scope of the study in Paris Region.
* Since informal caregivers can be included in the study by being linked to a previously included patient, the patient must agree to share the status with informal caregiver, or have previously shared their status with informal caregiver.
* Patients with legal protection may participate only if:
* They clearly agree that their legal representative should be consulted on participation in the study,
* They accept that this person is aware of their HIV status ,
* After having been consulted, this person (legally responsible) does not object to the participation of the person for whom he is responsible.

For informal caregiver:

* Person having a caring activity, before and during the study (such as the spouse, a child, a parent, neighbor, support person, etc.), for his close patient participating in the study,
* Authorized by the patient to be offered the study; the patient's agreement to approach the informal caregiver will have been sought beforehand in order to prevent the lack of medical confidentiality,
* Person expressing orally his non-opposition to his participation in the study and documented in the medical file of the patient to whom he is helping,
* Person capable of understanding the questionnaires and assessments of the study and able to answer them without the assistance of a third party.

For health professionals :

* Professional (health worker, nurse, coordinating physician, or other professions listed in the protocol), male or female, working in one of the study establishments recruited in Île-de-France (Nursing Home, Nurses home care services or Long-term care facilities), welcoming or having received people living with the Human Immunodeficiency Virus (HIV) ,
* Professional volunteer to participate in the study after having been informed with the information note intended for healthcare professionals.

Exclusion Criteria:

For patients:

* Patient expressing his opposition to his participation in the study,
* Patient who - according to the investigator - is unable to understand the study or answer the study questionnaires,
* Patient with a legal protection measure (guardianship and others), and at least 1 of the inclusion criteria for patients is not met.

For informal caregivers:

* Person not having a helping activity or exercising his role of helping for remuneration, or exercising his role of helping a loved one not included in the study,
* Person who exercises his role of helping in the context of a voluntary or associative activity,
* Person expressing orally his opposition to his participation in the study and documented in the medical file of the patient to whom he is helping,
* Person unable to understand the questionnaires and evaluations of the study and who is not able to answer them without the help of a third party,
* Person having the status of legal representative of the patient as part of a legal protection measure (guardianship and others).

For health professionals :

* Health professional working in the non-Francilians health or medico-social sector,
* Health professional opposing participation in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-positive patients in Paris region medico-social sector, their informal caregivers and health professionals in the medico-social sector.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The number of past situations for the last 5 years before the implementation of the study - of elderly people living with HIV in Retirement Home (EHPAD), home nursing care departments (SSIAD) and extended care units (USLD) in Île-de-France. | 2 years
The number of current situations for the last 5 years before the implementation of the study - of elderly people living with HIV in Retirement Home (EHPAD), home nursing care departments (SSIAD) and extended care units (USLD) in Île-de-France. | 2 years

SECONDARY OUTCOMES:
Assessment of the degree of patient dependence according "Index of Independence in Activities of Daily Living" KATZ scale | 2 years
  This is a measurement of the subject's ability to perform activities of daily living independently. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. A high score (6) indicates full function (patient independent). 2 or less score, indicates severe functional impairment.(patient very dependent)
Assessment of patient's level of dependence through an appreciation of instrumental activities of daily living according Lawton scale | 2 years
  The measure is calculated by summing the point values for each question. The maximum score of 8 indicates that all activities can be performed independently. A minimum score of 0 indicates that the measured activites of daily living can only be performed partially or not at all.
Assessment of depression according MINI Geriatric depression scale (Mini-GDS) | 2 years
  If the score is greater than or equal to 1: high probability of depression. If the score is 0: high probability of no depression.
Screening for undernutrition using Mini Nutritional Assessment (MNA) | 2 years
Assessment of quality of life according WHOQOL-HIV-BREF SCORE | 2 years
Measuring cognitive impairment according Mini-Mental State Examination (MMSE) score | 2 years
  The maximum score for the MMSE is 30. A score of 25 or higher is classed as normal. If the score is below 25, the result is usually considered to be abnormal (indicating possible cognitive impairment).
Assessment of somatic-comorbidities according Charlson scale | 2 years
Assessment of the degree of autonomy according AGGIR score | 2 years
Assessment of level of fargility according FREAD scale | 2 years
  5 is the best value, 0 is the worst value
Assessment of the emotional, physical and financial burden on a caregiver according Zarit burden scale | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hanon, MD PhD, Study Chair — Geriatric Department, Broca hospital,
Locations (1):
- Geriatric Department, Broca hospital, Paris, IIe-de-France, France